CLINICAL TRIAL: NCT01858129
Title: Inhaled Corticosteroids for the Treatment of Transient Tachypnea of the Newborn in Infants Born at >34 Weeks Gestation: A Prospective, Randomized, Double Blind, Placebo Controlled Study.
Brief Title: Inhaled Corticosteroids for the Treatment of Transient Tachypnea of the Newborn
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Bnai Zion Medical Center (Other Government)
Responsible Party: Principal Investigator, Kugelman Amir, Head, Pediatric Pulmonary Unit, Bnai Zion Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 0090-11-BNZ
Record Dates: First submitted 2013-05-14; First posted 2013-05-21 (Estimated); Last update posted 2015-01-29 (Estimated); Status verified 2015-01

CONDITIONS: Transient Tachypnea of the Newborn
Keywords: TTN
MeSH Terms: conditions — Transient Tachypnea of the Newborn

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Inhaled steroids (Budicort) (Experimental): Inhaled Budicort
  Interventions: Drug: Experimental group: Budicort by Inhalation
- Control (Placebo Comparator): Inhaled NS 0.9%
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: Experimental group: Budicort by Inhalation — Inhaled Budicort twice daily
  Arms: Inhaled steroids (Budicort)
Drug: placebo
  Arms: Control

SUMMARY:
Transient Tachypnea of the Newborn (TTN) is a common respiratory disorder affecting late preterm and term babies caused by lung edema resulting from delayed absorption of fetal alveolar lung fluid.

The investigators hypothesize that ENAC expression will be up-regulated as a result of administration of corticosteroids. This effect will lead to enhanced absorption of fetal lung fluid finally treating TTN. The aim of our study will be to evaluate whether inhaled corticosteroids reduce respiratory distress and morbidity in late preterm and term neonates presenting with TTN.

DETAILED DESCRIPTION:
The primary outcome measure will be the assessment of respiratory distress reflected by TTN clinical score in neonates presenting with TTN and treated with inhaled corticosteroids compared to placebo.

ELIGIBILITY:
Inclusion Criteria:

* Late preterm and term infants (post-menstrual age ≥ 34 weeks) delivered by cesarean section or vaginal delivery
* Diagnosis of TTN
* Parents signed informed consent

Exclusion Criteria:

* Meconium aspiration syndrome
* Respiratory distress syndrome
* Congenital heart disease
* Non respiratory disorders causing tachypnea

Ages: 4 Hours to 6 Hours | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 56 (Estimated)
Dates: Start 2012-03; Primary Completion 2015-05 (Estimated)

PRIMARY OUTCOMES:
Assessment of respiratory distress | 48 hours
  The primary outcome measure will be the assessment of respiratory distress reflected by TTN clinical score in neonates presenting with TTN and treated with inhaled corticosteroids compared to placebo at 12, 24 and 48 hours after the first dose of inhaled study medication.

SECONDARY OUTCOMES:
The secondary outcome will be the assessment of morbidity associated with TTN | An average time period expected to be 5 days, according to the duration of hospital stay
  The secondary outcome will be the assessment of morbidity associated with TTN as reflected by time to spontaneous unsupported breathing of room air (hours), time to spontaneous breathing (LFNC and/or FiO2<0.3) for infants who got a higher level of respiratory support, maximal level of respiratory support (no oxygen, intra-incubator oxygen, LFNC, nCPAP, NIPPV, high flow nasal canulla, SIMV, HFOV), LOS (days), TFF (hours), need and length of antibiotic therapy in the study vs. placebo groups.

OTHER OUTCOMES:
Will follow blood pressure | An average time period expected to be 5 days, according to the duration of hospital stay
  Blood pressure measurements

CONTACTS AND LOCATIONS:
Overall Officials: Amir Kugelman, MD, Principal Investigator — Bnai Zion Medical Center
Locations (1):
- Bnai Zion Medical Center, Haifa, Israel

REFERENCES:
- [Derived] Vaisbourd Y, Abu-Raya B, Zangen S, Arnon S, Riskin A, Shoris I, Elias N, Bader D, Kugelman A. Inhaled corticosteroids in transient tachypnea of the newborn: A randomized, placebo-controlled study. Pediatr Pulmonol. 2017 Aug;52(8):1043-1050. doi: 10.1002/ppul.23756. Epub 2017 Jul 3. PMID 28672098